### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

MEDICAL RECORD

Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 07-C-0059 PRINCIPAL INVESTIGATOR: William L. Dahut, M.D.

STUDY TITLE: A Phase II Study of AZD2171 in Metastatic Androgen Independent Prostate Cancer

Continuing Review Approved by the IRB on 7/20/09 Amendment Approved by the IRB on 12/4/09 (H)

Standard

Date Posted to the Web: 12/18/09

### INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health, (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical peliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

This is a clinical trial, a type of research study. Your study team will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to make your decision about taking part. You may discuss your decision with your friends and family or your referring physician. You can also discuss it with your study team. If you have any questions, you can ask your study doctor for more explanation.

You are being asked to take part in this study because you have a cancer that has not responded to standard treatments or for which no standard treatments have been identified.

PATIENT IDENTIFICATION

# CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (7-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent (1)

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

### **Description of Research Study**

### Why is this study being done?

The purpose of this study is to determine what effects, good and/or bad AZD2171, an unproven anticancer drug, has on you and your prostate cancer. This study will also help to determine how AZD2171 works in patients who have prostate cancer. AZD2171 is an experimental drug, not yet approved by the Food and Drug Administration. This study is being done in collaboration with Astra Zeneca, the makers of AZD2171, in an effort to understand the utility of this drug. The drug is an oral inhibitor of angiogenesis, the process of creating new blood vessels. All solid tumors require new blood vessels to grow. We hope to inhibit tumor growth with AZD2171 by preventing the growth of new blood vessels.

### How many people will take part in the study?

About 23 people will take part in this study.

What will happen if you take part in this research study?

This drug is a medicine you take by mouth and give to yourself every day. You will start by taking 1 tablet once daily. You are to swallow the tablet whole with about 8 oz. of water each morning, on an empty stomach, one hour before or two hours after meals. You should record the number of pills you consume and the time of consumption in a diary which will be provided to you by your study team. If you miss doses, that should also be recorded in the diary. If you remember your missed dose within three hours of the time you usually take a dose you may take a pill to make up for the missed dose; otherwise do not make up the missed dose. The dose will be adjusted if you experience any significant problems. This will be determined by your study team. AZD2171 can be taken while you are an outpatient. To help us to understand how the drug is working, a number of tests will be done, including tests to determine the level of vascular endothelial growth factor receptor (VEGFR), the target of AZDXIXI, in your blood prior to cycle 1 and monthly thereafter, as well as a special type of MRI (dynamic contrast-enhanced MRI, DCE-MRI, lasting approximately one hour) to evaluate blood flow, and tumor biopsies (optional), both before and after 2 and 6 cycles of treatment. You will be watched very closely as an outpatient and every 4 weeks return to the NIH to see a doctor who will monitor your response to the experimental treatment. At the outset of the study you may be hospitalized for 24 to 48 hours to complete research studies including your biopsies and blood measurements to determine the level of drug in your bloodstream. During this hospitalization, blood will be drawn immediatem prior to your first dose, and 0.25 hr, 0.5 hr, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, and 48 hours after ingestion. You will also have blood drawn at each clinic visit to measure the level of drug in your body. Each blood draw will consist of approximately one tablespoon of blood. In addition, you will be asked to take your blood pressure twice daily (once in the morning while resting quietly, once in the evening) and record it in a log which will be provided to you. Furthermore, all study participants will be invited to provide a blood sample (approximately one tablespoon) for retrospective evaluation of genetic variants possibly playing a role in how the drug acts. Participation in pharmacogenetic studies will be optional for all patients entering the study.

In addition, you will also take prednisone 10 mg per day. This drug is prescribed with FDA approved prostate cancer regimens. Our experience with this drug as well as at other institutions in individual patients demonstrates a possible benefit in decreasing some of the side effects from AZD-2171. At our institution, we have had four patients who have tried this combination and may have tolerated the AZD2171 better.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

### Before you begin the study ...

You will need to have the following exams, tests, and procedures to find out if it is safe for you to be in the study. The exams, tests, and procedures are part of regular cancer care and may be done even if you do not join the study. If you recently had some of the tests, they may not need to be repeated. This will be up to your study team.

- Blood tests: measurements of how your liver and kidneys work, measurement of your white blood cells, red blood cells and platelets, your blood sugar and blood electrolytes.
- Computerized Tomography scan of the chest, abdomen, and pelvis within the past 4 weeks
- Bone scan within the past 4 weeks
- Chest x-ray within the past 4 weeks
- Blood counts and chemistries (within 16 days before enrollment)
- PSA (Prostate Specific Antigen); if PSA is less than 4 ng/ml: PAP (prostate acid phosphatase) within 7 days of enrollment
- Tumor biopsy (optional)
- Electrocardiogram
- Echocardiogram

### During the study ...

If the exams, tests and procedures show that you can be in the study, and you shoose to take part, then you will need the following tests and procedures. Some are part of regular carcer care; other tests are specific to the drug you will be taking.

Blood tests including blood counts, chemistries, Thyroid Stimulating Hormone, and serum troponin.

- Electrocardiogram
- PSA measurements
- Urinalysis for protein.

You will need these tests and procedures that are also part of regular cancer care. They are being done more often because you are in this study.

- Computerized Tomography scan of the chest, abdomen, and pelvis and Echocardiogram after cycles 2 and 4, then every 3 months.
- Bone scan after cycles 2 and 4 ther every 3 months.

You will need these tests and procedures that are either being tested in this study or being done to see how the study drug is affecting your body.

- Pharmacokinetic sampling- this is determination of the amount of AZD2171 in your bloodstream at different amounts of time after having consumed the drug by mouth.
- Optional tumor biopsies before AZD2171 and after 2 and 6 cycles of experimental treatment.

Continue to record all doses of AZD2171 taken and / or missed in your pill diary. Record your blood pressure at least once daily in a blood pressure diary, which will be provided to you. We will also provide you with a blood pressure monitor.

### When you are finished taking AZD2171

Your participation in this study will continue until either you or your study team decides that this medication is not beneficial to you. Your participation is voluntary; so you may stop taking AZD2171 at any time, but we ask that you speak to your study team before stopping the study drug. Your study team will be monitoring you and your cancer while

NIH-2514-1 (10-84) NIH-2514-2 (10-84) P.A.: 09-25-0099

### **MEDICAL RECORD**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

you are taking AZD2171. If your prostate cancer is clearly worsening, then your study team will stop treatment with AZD2171. At the end of the study, no additional testing will be required.

### **Study Chart**

The treatment is given over 28-day periods of time called cycles. The 28 day treatment cycle will be repeated as long as you are tolerating the AZD2171 and your cancer is either steady or getting better. Each cycle is numbered in consecutive order. The chart below shows what will happen to you during Cycle 1 and future cycles. The left-hand column shows the day in the cycle and the right-hand column tells you what will happen on that day. This schedule indicates what will happen to you after you sign consent and start the study.

| | 976.6 = |
|---|---|
| Day | What to do and what will happen to you |
| Before | Get routine blood tests. |
| starting | Provide a history of how you feel and undergo a physical examination by a Health Care Provider. |
| AZD2171 | Research blood samples will be taken. |
| | Optional tumor biopsy (if there is a site that is safe as determined by your study team). You may |
| | require overnight admission to the hospital for the biogsy, the decision whether to admit will be |
| | discussed with you by your heath care team. |
| Day 1 | Begin taking AZD2171 once a day, and continue inless told to stop by your health care team. |
| | <ul> <li>Blood draws for research will be obtained on days 1 and 2 including a series of blood draws at</li> </ul> |
| | pre, 0.25 hr, 0.5 hr, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, and 48 hr after drug administration |
| | to monitor the level of AZD2171 in your bloodstream. You may be hospitalized overnight for |
| | these blood tests. |
| Day 2 | Do not take AZD2171 on Day 2 (because of the blood draws described above). |
| | Obtain weekly blood pressure checks at a healthcare facility. |
| | Check your blood pressure at home twice daily (once in the morning while resting quietly, and once |
| | in the evening) for the next 27 days. |
| | If you were admitted for biossies and other testing, you will be discharged from the hospital. |
| Day 3 | Bring AZD2171. Begin taking arog after your 48-hour blood draw. |
| Day 29 | Get routine blood tests and exams including PSA measurement. |
| (also Cycle | Return to the NIH clinic (OP)2 outpatient clinic) to see your doctor. Provide a history of how you feel |
| 2 day 1) | and undergo a physical examination by a Health Care Provider. |
| ' ' | If you are tolerating the drug well, the first dose of cycle 2 will be given at the NIH Clinical Center. |

### **Future cycles**

| Day | What to do and what will happen to you |
|---|---|
| Days 1-28 | Keep taking AZD2171 once a day if you have no bad side effects and cancer is not getting worse. |
| | Call the research nurse, , or your study doctor if you do not know what to do. |
| | Get routine X-rays, |
| | Computerized Tomography scans, Echocardiograms and/or bone scan cycles 2 and 4, then |
| | every 3 months (more if your doctor tells you to). |
| | MRIs cycles 2 and 4, then every 4 months |
| | Optional tumor biopsy after cycles 2 and 6; biopsy may require overnight admission. |
| Day 29 | Return to your doctor's office for your next exam and to begin the next cycle. |

NIH-2514-1 (10-84) NIH-2514-2 (10-84) P.A.: 09-25-0099

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

### How long will you be in the study?

You will be invited to continue to take AZD2171 until your study team advises you that the medication is not helping your cancer, you are experiencing significant toxicity from the therapy, or you decide that you no longer wish to participate in the study.

### Can I stop being in the study?

Yes. You can decide to stop at any time. Tell your study team if you are thinking about stopping or decide to stop. He or she will tell you how to stop safely.

It is important to tell your study team if you are thinking about stopping so any risks from AZD2171 can be evaluated by your study team. Another reason to tell your study team that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

Your study team may stop you from taking part in this study at any time if they believe it is in your best interest, if you do not follow the study rules, or if the study is stopped.

### **Alternative Approaches or Treatments**

### What other choices do I have if I do not take part in this study?

To make an informed decision about whether or not to participate in this study, you need to know your options. Alternative treatments to this study, in general, include:

- 1) no further treatment of the cancer, but treatment of any symptoms that may be causing discomfort, this type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.
- 2) chemotherapy and/or hormonal therapy with commercially available drugs. Recent studies have shown that a drug known as docetaxel or taxotere in combination with prednisone has survival benefit in prostate cancer. This is now recognized as the standard treatment of prostate cancers that are no longer sensitive to hormonal therapies. You are required to have at least one attempt at cytotoxic therapy for your prostate cancer before enrolling on this study; you remain eligible for this study after several attempts at different types of cytotoxic therapy.
- 3) ketoconazole
- 4) other experimental therapies,
- 5) radiation therapy to shrink tumor masses or relieve pain, and
- 6) surgery to remove tumor masses.

All of these options may not apply to your particular situation, but it is important that you have explored these options with your regular doctor.

### **Risk or Discomforts of Participation**

### What side effects or risks can you expect from being in the study?

You may have side effects while you are taking the study drug. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen so it is important to report changes that you may notice, even if your study team does not ask specifically about them. Side effects may be mild or very serious. Your study team may give you medicines to help lessen side effects. Many side effects go away with those medicines and others can go away soon after you stop taking AZD2171. In some cases, side effects can be

### **MEDICAL RECORD**

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059

CONTINUATION:  pages

serious, long lasting, or may never go away. There are no known long-lasting toxicities from AZD2171 at this time. You should talk to your study team about all side effects that you have while taking part in the study.

Preliminary studies have shown hypertension, or elevated blood pressure, to be one common side effect of AZD2171. Your blood pressure will be closely monitored while you are taking AZD2171. If your blood pressure becomes elevated while taking AZD2171, your physicians may recommend follow-up with your primary care physician, starting or increasing medication to lower blood pressure, and / or home blood pressure monitoring.

Grapefruit juice has been shown to interact with a number of drugs by blocking the activity of the body's cytochrome P450 (CYP450) system. CYP450 is important in breaking down substances in the body, including many drugs. Since the degree to which grapefruit juice interacts with AZD2171 in the body is not fully known, please avoid grapefruit juice while taking AZD2171. As other drugs may also interact with the CYP450 system, please contact the study team prior to starting any new medication.

Risks and side effects related to AZD2171 are detailed in the table on the following page. "Common" side effects as those occurring in greater than 20% of patients and "Uncommon" side effects as those occurring in  $\leq$  20% of patients.

Risks and side effects related to AZD2171 include those which are:

| Side Effect | Mild | Severe, but not life threatening | Life threatening |
|---|---|---|---|
| Common | High blood pressure (Hypertension) Diarrhea (can be severe in some cases) Fatigue Loss of appetite (Anorexia) Hoarseness, loss or alteration in voice, throat irritation | | |
| Uncommon | (laryngitis) Red peeling rash affecting the hands and feet (hand-foot syndrome) Abnormal blood tests related to liver function Dry mouth Headache (can be severe in some cases) Constipation Weight loss Cough Sweating Low thyroid function (with associated inreased thyroid stimulating hormone | | |

### **MEDICAL RECORD**

#### **CONTINUATION SHEET for either:**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

| | and decreased thyroxine levels) Dehydration Proteinuria (protein in the urine) Difficulty swallowing (dysphagia) Mouth ulcers (mucositis) Muscle pain Fever , Back pain, Joint pain, Muscle pain Nausea Vomiting Shortness of breath Dry Skin Abdominal Pain Decreased platelets Bladder spasms Low red blood cells causing anemia Low blood pressure | | |
|---|---|---|---|
| Rare | Hypokalemia* | Duodenal ucer (stomach ulcer)* Aphasia (inachlity to speak)* Hepatic heriotrhage (bleeding into the liver)* Abnormal EKO (prolonged QT corrected)* Muscle weakness* Transient ischemic attack ("ministroke")* Deer vein thrombosis (blood clots)* Left ventricular systolic dysfunction (decrease in heart function) Formation or presence of a blood clot inside an artery Leukoencephalopathy syndrome including reversible posterior leukoencephalopathy syndrome (RPLS). RPLS is a medical condition related to leakiness of blood vessels in the brain and can cause confusion, blindness or vision changes, seizure and other symptoms, as well as changes in brain scans. This condition is usually reversible, but in rare cases it is potentially life-threatening and may have long-term effect on brain function. | Low blood sugar* Stroke* Hypertensive crisis (severe high blood pressure) Lung infection/pneumonia* Bleeding into you spine or brain(Central Nervous System Hemorrhage)* Death* Kidney Failure(Renal Failure)* |

<sup>\*</sup>Duodenal ulcer (stomach ulcer), Hepatic hemorrhage (bleeding into the liver), transient ischemic attack (ministroke), deep vein thrombosis (blood clots), low blood sugar, abnormal EKG (prolonged QT corrected), muscle weakness, aphasia (inability to speak), Low Potassium (Hypokalemia), Lung infection/pneumonia, Bleeding into you spine or brain(Central Nervous System Hemorrhage)\*, Death, Kidney Failure (Renal Failure) and stroke are classified as rare side effects of

#### **MEDICAL RECORD**

NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

AZD2171. These events have occurred on AZD2171 trials but it has not yet been determined whether the events were caused by AZD2171.

Reproductive risks: You should not father a baby while on this study because the drugs in this study can affect an unborn baby. It is important you understand that you must refrain from intercourse or need to use birth control while on this study. Check with your study doctor about what kind of birth control methods to use and for how long you should use them after you are no longer receiving the study drug. Typical birth control methods include abstinence from intercourse, barrier contraceptives (condoms, diaphragms), or hormonal agents (oral contraceptive pills).

For more information about risks and side effects, ask your study team.

AZD2171 can cause hypertension that can become significant. For the first 4 weeks of the study you will be required to have your blood pressure checked at a healthcare facility. This should be recorded in your first study diary and reported to the research team.

You will also begin taking prednisone by mouth at a dose of 10 mg on the first tax of each cycle but you will continue to take it daily throughout the cycle. The side effects that have been associated with prednisone include:

- •gastric hyperacidity(increased stomach acid), increased appetite, insorbina or nervousness occurring in > 10% of patients
- •hyperglycemia (high blood sugar level), fluid retention, mood swings, dizziness, headaches, muscle weakness, osteoporosis (bone thinning), and cataracts with long-term use, occurring in about 1% 10% of patients

\*Hypertension occurring in < 1% of patients but this risk may be higher in combination with AZD2171.

In addition, this combination of prednisone and AZD-2271 has not been studied before so unknown side effects may also occur.

The DCE-MRI involves intravenous injection with a special non-radioactive dye (gadolinium chelate) to examine blood flow in a certain part of the body. An intravenous injection involves a needle stick into a vein in the arm. Several attempts may be necessary to place the needle into the vein. In addition to the pain associated with the needle stick there may be some bruising after the needle is removed. Experience with a large number of patients who have received commercially available gadolinium has shown it is without side effects in a large majority of patients. When side effects do occur, they are usually mild and last a short time. These include coolness in the arm during injection, headache, and nausea. More severe reactions (shortness of breath, wheezing, or lowering of blood pressure) have occurred in an extremely small number of patients.

Side effects may be mild or very serious. Many side effects go away soon after you stop taking AZD2171. In some cases side effects may be long lasting or may never go away. There also is a risk of death.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

### **Potential Benefit**

### Are there benefits to taking part in the study?

Taking part in this study may or may not make your health better. While doctors hope AZD2171 will be more useful against cancer compared to currently available treatments, there is not yet any proof that this is so. We do know that the information from this study will help doctors learn more about AZD2171 as a treatment for cancer. The information will help future cancer patients.

### Cost and Reimbursement

### What are the costs of taking part in this study?

While you are on study at the National Cancer Institute, we will pay for the medications and treatments associated with the study. We cannot, however, assume the cost of your overall medical care. Any studies done outside of the NCI may require you or your insurance company to cover the cost of the service.

You will not be paid for taking part in this study.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER/(1-800-422-6237) and ask them to send you a free copy.

## What happens if you injured because you took part in this study?

It is important that you tell your study team, Principal in this study. You will get medical treatment if you are injured as a direct result of taking part in this study at the NIH.

### What are your rights if you take part in this study?

Taking part in this study is your choice. You may choose either to take part or to not take part in the study. If you decide to take part in this study, you may be the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any or your regular benefits. You can still get your medical care from our institution if you are eligible and choose to participate in another trial.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

### Communication

### Who can answer my questions about the study?

You can talk to your study doctor about any questions or concerns you have about this study. Contact your study team (Principal Investigator Dr. William Dahut) at (301) 435-5613,

If you have any complications when you are not in the Clinical Center (e.g., at home or in a local hotel), you may call the page operator at (301) 496-1211 and ask for the NCI Medical Oncology Branch physician on call or the NIH Patients'

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

Rights Representative who will be available to answer questions concerning your involvement in this study or your rights as a research subject. She is not directly associated with this study and can be contacted at (301) 496-2626.

### Research Subjects' Rights

### Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- Qualified representatives from AstraZeneca Pharamceuticals, the pharmaceutical drug sponsors who produce AZD2171.

Please note: This section of the informed consent form is about additional studies that are being done with people who are taking part in the main study. You may take part in these additional studies if you want to. You can still be a part of the main study even if you say 'no' to taking part in any of these additional studies. You can say "yes" or "no" to each of the following studies. Please mark your choice for each study.

### **About Using Tissue for Research**

We encourage all patients on this study to agree to tumor biopsies for research purposes, at intervals as described in this consent. Participating in biopsies is optional; study enablidity is not contingent on agreeing to tumor biopsy. If you agree to biopises, your doctor will remove some body tissue do some tests. None of the data gained by the biopsy will affect your participation in the study. The intention of obtaining the tissue is solely scientific and will not be used to direct your care.

Reports about research done with your tissue will not be given to you or your doctor. These reports will not be put in your health record. The research will not have an effect on your care.

#### Things to Think About

If you decide now that your tissue can be kept for research, you can change your mind at any time. Just contact us and let us know that you do not want us to use your tissue. Then any tissue that remains will no longer be used for research.

In the future, people who do research may need to know more about your health. While the NCI may give them reports about your health, it will not give them your name, address, phone number, or any other information that will let the researchers know who you are.

Your tissue will be used only for research and will not be sold. The research done with your tissue may help to develop new products in the future.

### **Benefits**

The benefits of research using tissue include learning more about what causes cancer and other diseases, how to prevent them, and how to treat them.

**MEDICAL RECORD** 

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

#### **Risks**

The greatest risk to you is the release of information from your health records. We will do our best to make sure that your personal information will be kept private. The chance that this information will be given to someone else is very small.

### **Making Your Choice**

Please read each sentence below and think about your choice. After reading each sentence, circle "Yes" or "No". If you have any questions, please talk to your doctor or nurse, or call the NIH Clinical Center Patient Representative at (301) 496-2626. No matter what you decide to do, it will not affect your care.

1. My tissue may be kept for use in research to learn about, prevent, or treat cancer.

Yes No

2. My tissue may be kept for use in research to learn about, prevent or treat other health problems (for example: diabetes, Alzheimer's disease, or heart disease).

Yes No

3. Someone may contact me in the future to ask me to take part in more research

Yes

Where can I get more information?

You may call the National Cancer Institute's Cancer Information Service at: 1-800-4-CANCER (1-800-422-6237) or TTY: 1-800-332-8615

You may also visit the NCI Web site at http://cancer.gov

- For NCI's clinical trials information, go to http://tancer.gov/clinicaltrials/
- For NCI's general information about cancer, go to <a href="http://cancer.gov/cancerinfo/">http://cancer.gov/cancerinfo/</a>

You will get a copy of this form. If you want more information about this study, ask your study doctor.

NIH-2514-1 (10-84) NIH-2514-2 (10-84) P.A.: 09-25-0099

### **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY**

**MEDICAL RECORD** 

• Adult Patient or • Parent, for Minor Patient

STUDY NUMBER: 07-C-0059 CONTINUATION:  pages

### OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- **2. Policy Regarding Research-Related Injuries.** The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, William L. Dahut, M.D. at (301) 435-5613; Building 10, Room 12N226.

You may also call the Clinical Center Patient Representative at 301-496-2626.

5. Consent Document. Please keep a copy of this document in case you want to read it again.

| COMPLETE APPROPRIATE YTEM(S) BELOW: | | |
|---|---|---|
| A. Adult Patient's Consent I have read the explanation about this study and have been given opportunity to discuss it and to ask questions. I hereby consent to be part in this study. | <b>B.</b> Parent's Permission for Minor Patient. I have read the explanation about this study and have been given the | |
| Signature of Adult Patient/Legal Representative Date | Signature of Parent(s)/Guardian Date | _ |
| Print Name | Print Name | |
| C. Child's Verbal Assent (If Applicable) The information in the above consent was described to my child and my child agrees to participate in the study. | | |
| Signature of Parent(s)/Guardian Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM JULY 20, 2009 THROUGH JULY 19, 2010. | | |
| Signature of Investigator Date | Signature of Witness Date | |
| Print Name | Print Name | |

### **PATIENT IDENTIFICATION**

CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or • Parent, for Minor Patient

NIH-2514-1 (7-09)

P.A.: 09-25-0099 File in Section 4: Protocol Consent FAX TO: (301) 480-3126